CLINICAL TRIAL: NCT02909803
Title: Measuring the Glycemic Index and Tracking Metabolites of New and Emerging Lentil Varieties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guelph Food Research Centre (Other Government)
Collaborators: Glycemic Index Laboratories, Inc (Industry); University of Manitoba (Other)
Responsible Party: Principal Investigator, Dan Ramdath, Research Scientist, Guelph Food Research Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Lentil metabolites
Record Dates: First submitted 2016-09-15; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Hyperglycemia; Dietary Modification
Keywords: glucose; glycemic index; lentil; polyphenols; metabolites; bioavailability
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lentil Variety (Experimental): Each participant will consume a serving of one of eight lentil varieties (Greenland; Improve; Impower; Imigreen; Asterix; Redberry; Redcliff; Redbow) containing 25g available carbohydrate at separate study visits
  Interventions: Other: Lentil Variety
- White Bread (Active Comparator): Each participant will consume a serving of white bread containing 25g available carbohydrate on two separate visits
  Interventions: Other: White Bread

INTERVENTIONS:
Other: Lentil Variety — Participants will consume 8 varieties of lentils that are cooked by boiling
  Arms: Lentil Variety
Other: White Bread — Participants will consume white bread on at least two different test days
  Arms: White Bread

SUMMARY:
It is not known whether different lentil varieties have the same efficacy in lowering blood glucose. Similarly, the carbohydrate component of lentils responsible for lowering blood glucose is not known, nor is the bioavailability of lentil metabolites and polyphenol bioactive.

DETAILED DESCRIPTION:
The overall aim of this work is to produce credible evidence for substantiating a food health claim for post prandial blood glucose lowering by lentil. Although several studies have shown that lentil consumption results in a lowering of post prandial blood glucose, it is not known whether different lentil varieties have the same efficacy. Similarly, the carbohydrate component of lentils responsible for lowering blood glucose is not known, nor is the bioavailability of lentil metabolites and polyphenol bioactive. The investigators hypothesize that the slowly digestible starch content of lentil is inversely related to in vivo glycemic response. The specific aims of this study are: (i) to identify the putative component(s) in lentil that might account for its blood glucose lowering effect, and (ii) to identify differences in blood glucose reduction among lentil varieties. These aims will be achieved in a three-step process. Firstly, in vitro studies will be pursued to determine the carbohydrate fractions of 20 new and emerging Canadian lentil varieties. Secondly, these results will be used to choose 8 lentil varieties with different slowly digestible starch content for a human Glycemic Index study. Thirdly, identification of lentil metabolites will be achieved by collecting extra capillary blood (200uL)and urine samples at fasting and 120min for measurement of polyphenols and metabolites using established HPLC and metabolomics techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-75 years of age, inclusive
* Body mass index (BMI) < 40 kg/m²
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, diabetes or a heart condition
* Subjects using medications or with any condition which might, in the opinion of Dr. Wolever, the Medical Director of GI Labs, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Glycemic Response | 120 minutes after consuming each test or control food
  Incremental blood glucose response after eating the test or control foods will be measured over a period of 120 minutes using finger prick blood samples collected at time 0, 15, 30, 45, 60, 90, 120 minutes.

SECONDARY OUTCOMES:
Lentil metabolites in blood and urine | Urine and additional 200uL blood samples will be collected before eating test meal and at 120 minutes after.
  Samples will be preserved and analyzed for polyphenols (HPLC) and unknown metabolites using a non-targeted metabolomics approach.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ramdath, PhD, Principal Investigator — Guelph Research and Development Centre
Locations (1):
- Glycemic Index Laboratories, Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Health Canada. Bureau of Nutritional Sciences, food directorate, health products and food branch. June 2013. Draft guidance document on food health claims related to the reduction in post-prandial glycaemic response
- [Background] Wolever TM, Jenkins DJ. The use of the glycemic index in predicting the blood glucose response to mixed meals. Am J Clin Nutr. 1986 Jan;43(1):167-72. doi: 10.1093/ajcn/43.1.167. PMID 3942088
- [Background] Wolever TMS (2006). The Glycaemic Index: A Physiological Classification of Dietary Carbohydrate. CABI Publishing, Wallingford, UK.
- [Background] Ramdath D, Renwick S, Duncan AM. The Role of Pulses in the Dietary Management of Diabetes. Can J Diabetes. 2016 Aug;40(4):355-63. doi: 10.1016/j.jcjd.2016.05.015. PMID 27497151
- [Background] Wang, L., Zahradka, P., Taylor, C. and Aliani, M., Metabolomics Analysis of Serum and Urine After Bean Consumption by Patients with Peripheral Arterial Disease. The FASEB Journal, 30(1 Supplement): 682-10, 2016.